CLINICAL TRIAL: NCT03124758
Title: Accuracy of Noninvasive Hemoglobin Sensor (Rainbow Reusable DCI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TR24577-TP15879-TP14065
Record Dates: First submitted 2017-04-14; First posted 2017-04-24 (Actual); Results first posted 2017-06-06 (Actual); Last update posted 2017-07-27 (Actual); Status verified 2017-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Noninvasive Hemoglobin Sensor (Experimental): All subjects are enrolled into the test group and all subjects received the Noninvasive Hemoglobin Sensor (Rainbow Reusable DCI, DCIP)
  Interventions: Device: Hemoglobin Sensor ((Rainbow Reusable DCI, DCIP))

INTERVENTIONS:
Device: Hemoglobin Sensor ((Rainbow Reusable DCI, DCIP)) — Measurement of Noninvasive Hemoglobin (SpHb)

SUMMARY:
In this study, the accuracy of a noninvasive hemoglobin sensor(s) will be assessed by comparison to hemoglobin measurements from a laboratory hematology analyzer. Blood samples are collected from healthy volunteers who are enrolled in either a blood draw procedure or a hemodilution procedure wherein blood is repeatedly sampled as the concentration of hemoglobin is reduced in a controlled manner by administering fluids intravenously.

ELIGIBILITY:
A. Hemodilution Test Procedure

Inclusion Criteria:

* Weight of more than 110 lbs and less than 220 lbs.
* Physical status of ASA I of II
* Able to read and communicate in English
* Has signed written informed consent
* Female, non pregnant. Female subjects will be provided with a pregnancy test free of charge.

Exclusion Criteria

* Age less than 18 yrs and greater than 35 years
* Weight of less than 110 lbs or more than 220 lbs.
* Hemoglobin less than 12 g/dL
* ASA physical status of III. IV, V.
* Pregnant
* Subject has known drug or alcohol abuse
* Subject has skin abnormalities affecting the digits such as psoriasis, eczema, angioma, scar tissue, burn, fungal infection, substantial skin breakdown, nail polish or acrylic nails.
* Subject has experienced a head injury with loss of consciousness within the last year
* Subject has known neurological and psychiatric disorder that interferes with the subjects level of consciousness
* Known or concurrent chronic usage of psychoactive or anticonvulsive drugs within the last 90 days, or any use in the last 7 day (i.e. tricyclic antidepressants, MAO inhibitors, Lithum, neuroleptics, anxiolytics or antipsychotics, except SSRIs).
* Subject has any medical condition which in the judgment of the investigator, renders them inappropriate for participation in this study, such as Reynauds Syndrome.
* Hypertension: Systolic BP >140 mmHg or Diastolic BP > 90 mmHg.
* Baseline heart rate < 50 bpm.
* Inability to tolerate sitting still or minimal movement for up to 90 minutes
* Discretion of investigator

B. Blood Draw Test Procedure

Inclusion Criteria:

-Subjects must understand and consent to be in the study.

Exclusion Criteria

* Subjects less than 18 years of age.
* Subjects who do not understand the study and the risks involved.
* Anyone deemed ineligible by test personnel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 354 (Actual)
Dates: Start 2010-04-20 (Actual); Primary Completion 2011-10-31 (Actual); Study Completion 2011-10-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Masimo Corporation, Irvine, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Noninvasive Hemoglobin Sensor
Started | 354
Completed | 354
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Noninvasive Hemoglobin Sensor
Number analyzed (Participants) | 354
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 354
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127
  Male | 227

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of Sensor by Arms Calculation
Description: Accuracy will be determined by comparing the noninvasive hemoglobin measurement of the pulse oximeter to the hemoglobin value obtained from a blood sample and calculating the arithmetic root mean square(Arms) error value.
Time Frame: 1-5 hours
Measure: Number; unit: g/dL
Units Other Than Participants: data points
Arm/Group | Noninvasive Hemoglobin Sensor
Number analyzed (Participants) | 354
Number analyzed (data points) | 1990
g/dL | 1.0

ADVERSE EVENTS:
Arm/Group | Noninvasive Hemoglobin Sensor
Serious Adverse Events (participants affected / at risk) | 0/354
Other Adverse Events (participants affected / at risk) | 0/354

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes